CLINICAL TRIAL: NCT06200974
Title: Multi-omic Approach to Study High Dose Rate (HDR) Brachytherapy for Favorable Risk and Low Tier Intermediate Risk Prostate Cancer
Brief Title: Multi-omic Approach to Study HDR Brachytherapy for Favorable Risk and Low Tier Intermediate Risk Prostate Cancer
Acronym: BrachyTRACKS
Status: Recruiting | Type: Observational
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: BC Cancer Foundation (Other); University of British Columbia (Other); Vancouver Prostate Centre (Other)
Responsible Party: Principal Investigator, Juanita Crook, Professor of Radiation Oncology, British Columbia Cancer Agency
Other Study IDs: H23-02872
Record Dates: First submitted 2023-12-13; First posted 2024-01-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Localized Prostate Carcinoma
Keywords: Brachytherapy; TRACKS; High Dose Rate; Prostate cancer; favorable risk; intermediate risk
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High dose rate prostate brachytherapy: Radiation. High dose rate prostate brachytherapy is delivered under anesthesia in 2 procedures, 1-2 weeks apart.
  HDR brachytherapy is also accomplished as an out-patient.
  Interventions: Radiation: High dose rate prostate brachytherapy

INTERVENTIONS:
Radiation: High dose rate prostate brachytherapy — Temporary implantation of radioactive material into the prostate in the form of a stepping source of Iridium 192 that travels through 16-18 needles or catheters strategically placed through the prostate.
  Other Names: HDR brachytherapy

SUMMARY:
This is an observational single-center trial for patients with localized prostate cancer suitable for High Dose Rate (HDR) brachytherapy as monotherapy. This study takes a multi-omics approach to study the mechanism of action of HDR brachytherapy through metabolomics, immunological, transcriptomics, and spectroscopic profiling. The results of this study will clarify the optimal dose for HDR prostate brachytherapy by documenting the dose-response relationship seen in the changing tumor metabolites after HDR brachytherapy and investigate the immunogenicity of HDR brachytherapy.

DETAILED DESCRIPTION:
High Dose Rate (HDR) prostate brachytherapy is an effective and highly conformal means of delivering curative radiation to the prostate. Because of the high dose rate, initial studies applied this treatment cautiously in multiple sessions or fractions but this has gradually been reduced from 54 Gy in 9 fractions to 42 Gy in 6, then 36 Gy in 3, then 27 Gy in 2 and finally to one single fraction of 19 Gy. Each change in fractionation was calculated to be equivalent to the previous, and remarkably, efficacy was maintained until the final stage when treatment was reduced to a single fraction. This resulted in a significant drop in cure rates from over 90% to approximately 65%. The investigators assume that the prior fractions served to sensitize the tumor to subsequent radiation; however, this remains an open question.

This observational single-center trial for localized prostate cancer suitable for brachytherapy as monotherapy takes a novel multi-omics approach to study the mechanism of action of High Dose Rate (HDR) brachytherapy through metabolomics, immunological, transcriptomics, and spectroscopic profiling. This is achieved through (1) measurement of changes in metabolites as determined by Raman spectroscopy, (2) analysis of circulating tumor DNA in peripheral blood plasma, (3) evaluation of the changes in immune response by single cell RNA (scRNA)-sequencing, and (4) evaluation of gut microbiome composition before and after treatment. Secondary endpoints of the study include PSA nadir, time to nadir, PSA at 4 years and patterns of failure.

The study will enroll 100 men with localized prostate cancer suitable for brachytherapy as monotherapy. HDR brachytherapy is given in 2 fractions, each one under anesthesia, making it possible to obtain biopsies painlessly at both baseline prior to any treatment, and 1-2 weeks later prior to the second half of treatment. The results of this study will clarify the dose-response relationship for HDR brachytherapy, help to define the optimal dose, clarify the metabolic response to HDR brachytherapy, and investigate the potential immunogenicity of HDR brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* Favorable risk and intermediate-risk prostate cancer with estimated life expectancy of at least 10 years.
* Clinical stage T1c-T2b, PSA < 20, Gleason < 8
* ECOG 0-1
* Low tier intermediate-risk prostate cancer is defined by: a single NCCN intermediate risk factor (either Gleason 7(3+4) and PSA < 10 ng/ml OR Gleason 6 and PSA 10-20 ng/ml)
* Extensive favorable-risk disease is defined as: clinical stage T1c-T2a, PSA < 10, Gleason 6, ≥ 50% of biopsy cores containing cancer, PSA density > 0.2 ng/cc,
* Selected intermediate risk patients not defined above

  * T1c/T2a
  * PSA < 10 and Gleason 4+3
  * PSA > 10 (< 20) and Gleason 3+4
  * PSA 10-15 ng/ml and Gleason 4+3 and < 33% cores involved
  * Max tumor length in any core 10 mm
* No androgen deprivation therapy (ADT)
* Signed study specific informed consent.

Exclusion Criteria:

* Prior radical surgery for carcinoma of the prostate,
* Prior pelvic radiation
* Prior chemotherapy for prostate cancer,
* Claustrophobic or unable to undergo MRI
* Patients unsuitable for general anesthesia, on blood thinners which cannot be stopped for 24 hours, or who have contraindications to radiotherapy such as systemic sclerosis, or inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with localized prostate cancer suitable for brachytherapy as monotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2038-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in biomolecular composition in prostate cancer after high dose rate prostate brachytherapy as measured by Raman spectroscopy | 1-2 weeks, PSA: 0-10 years
  We will report the most important biomolecules altered by radiation (importance determined by the relative change of the score as a component of the Raman spectrum before and after radiation) and whether that observed change corelates with PSA outcome for each individual patient
ctDNA detection following HDR Brachytherapy | 0-4 weeks
  Number of patients with a (transient) increase in circulating tumor DNA after a single fraction of high-dose rate prostate brachytherapy will be reported
Immunogenicity against somatic mutations | 0-4 weeks
  single cell-RNA sequencing of immune cell populations before and after 13.5 Gray of radiation will be used for each individual patient and the number of patients with a change in gene expression (through activation or inactivation) will be reported
Gut microbiome | 0-4 weeks
  To determine microbial composition before brachytherapy and report for the individual patient whether diversity in composition is changed or skewed after treatment with high dose rate prostate brachytherapy. Second assessment is after completion of both fractions of radiation. Number of patients with alteration in microbial composition will be reported.

SECONDARY OUTCOMES:
Response Outcome: PSA Nadir | 0-10 years
  PSA recorded every 3 months to 12 months, every 6 months to 3 years, and annually to 10 years
Response Outcome: 4-year PSA | 0-4 years
  4-year PSA < 0.2 ng/ml (indicative of cure)
Acute and long term toxicity | 0-10 years
  Acute and long-term toxicity will be graded using the Common Terminology Criteria for Adverse Events (CTCAE V5) at each follow up time point

CONTACTS AND LOCATIONS:
Overall Officials: Juanita M Crook, MD, Principal Investigator — Radiation Oncologist
Locations (1):
- British Columbia Cancer Center for the Southern Interior, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No